CLINICAL TRIAL: NCT04439201
Title: MATCH Treatment Subprotocol Z1B: Phase II Study of Palbociclib (PD-0332991) in Patients With Tumors With CCND1, 2, 3 Amplification
Brief Title: Testing Palbociclib (PD-0332991) as a Potential Targeted Treatment in Cancers With CCND1, 2, 3 Amplification (MATCH-Subprotocol Z1B)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03171; NCI-2020-03171 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1B (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1B (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (palbociclib) (Experimental): Patients receive palbociclib PO QD days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991

SUMMARY:
This phase II MATCH treatment trial identifies the effects of palbociclib in patients whose cancer has genetic changes called CCND1, 2, or 3 amplification. Palbociclib blocks proteins called CDK4 and CDK6, which may stop cancer cell growth when CCND1, 2, or 3 amplifications are present. Researchers hope to learn if palbociclib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive palbociclib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have amplification of CCND1, 2, or 3, or another aberration, as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)

Exclusion Criteria:

* Patients must not have known hypersensitivity to palbociclib or compounds of similar chemical or biologic composition
* Patients must not have breast cancer, mantle cell lymphoma or myeloma
* Patients with known or symptoms of left ventricular dysfunction will be excluded
* Patients must not have had prior treatment with palbociclib, ribociclib, abemaciclib or any other CDK4/6 inhibitors
* Patients must not be using drugs or foods that are known potent CYP3A4 inhibitors or inducers, or are CYP3A4 substrates with narrow therapeutic indices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Clark, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1B was activated on May 31, 2016. Forty patients were enrolled between August 2016 and December 2017.
Pre-assignment Details: To be eligible for this subprotocol, tumors had to contain both an amplification in CCND1, 2, or 3 and Rb expression. CCND amplification was defined as seven or more copies of the gene; Rb expression was defined as 1+ or greater staining by IHC. The mutation status was determined by a CLIA-approved assay performed in a NCI-MATCH approved laboratory for all patients in this arm. Confirmatory central testing was required in order for these patients to be included in the primary analysis.
Groups:
- Treatment (Palbociclib): Patients receive palbociclib 125 mg PO QD days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Palbociclib: Given PO
Period: Overall Study
Arm/Group | Treatment (Palbociclib)
Started | 40
Eligible | 37
Started Protocol Therapy | 38
Eligible and Treated | 36
Mutation Status Confirmed | 36
Eligible, Treated and Mutation Status Confirmed (This is the primary analysis population.) | 32
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 40
Not completed — Ineligible | 2
Not completed — Never start protocol therapy | 1
Not completed — Ineligible and never start protocol therapy | 1
Not completed — Mutation status not confirmed | 4
Not completed — Adverse Event | 1
Not completed — Death | 7
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 20
Not completed — Alternative therapy | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 62 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 32
Participants | 0

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 32
percentage of participants | 16 [8 to 35]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 32
months | 1.8 [1.5 to 2.7]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-eight patients were included in the toxicity analysis (excluding two who did not receive treatment).
Arm/Group | Treatment (Palbociclib)
All-Cause Mortality (participants affected / at risk) | 38/40
Serious Adverse Events (participants affected / at risk) | 20/38
Other Adverse Events (participants affected / at risk) | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palbociclib) (N=38)
Anemia (Blood and lymphatic system disorders) | 2
Death NOS (General disorders) | 1
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palbociclib) (N=38)
Anemia (Blood and lymphatic system disorders) | 12
Fatigue (General disorders) | 9
Fever (General disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 13
Platelet count decreased (Investigations) | 11
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 17
Investigations - Other, specify (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04439201/Prot_001.pdf